CLINICAL TRIAL: NCT04426422
Title: Effect of Metformin on Gut Microbiota Changes and Glycemic Control of Newly Diagnosed Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUTT2DM
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: newly diagnosed type 2 diabetes was treated with metfomin for 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metformin group (Experimental): all the patients were treated with metformin 1500-2000mg daily for 3 months.
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — treated with metformin 1500-2000mg daily
  Other Names: intervention group

SUMMARY:
This study was aimed to investigate the effect of metformin on the gut microbiota and glycemic control in newly diagnosed type 2 diabetes patients.

DETAILED DESCRIPTION:
This study was aimed to investigate the effect of metformin on the gut microbiota and glycemic control in newly diagnosed type 2 diabetes patients. All the recurited patients were treated with metformin 1500-2000mg daily for 3 months. Stool specimens and blood samples were collected at the beginning and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

newly diagnosis type 2 diabetes ,HbA1c >7 %

Exclusion Criteria:

history of cardiovascular disease, hypertension, severe renal dysfunction defined as glomerular filtration rate < 45 mL/min/1.73 m2; severe illness or diabetic ketoacidosis within 30 days, inability to tolerate ≥500 mg metformin twice per day and pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
gut micribiota | 3 months
  the changes of gut micribiota

SECONDARY OUTCOMES:
glycemic control | 3 months
  HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: fengyi Yuan, Principal Investigator — Shenzhen People' hospital
Locations (1):
- Shenzhen People' S Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
no decided yet.